CLINICAL TRIAL: NCT02773927
Title: Effect of the Combination Metformin/Inulin vs Inulin on Adiponectin in Patients With Metabolic Syndrome
Brief Title: Combination of Metformin/Inulin vs Inulin on Adiponectin in Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Fernando Grover-Paez, PhD, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUCS-INTEC-MV-HBP-002
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Metabolic Syndrome
Keywords: Agave inulin; Adiponectin; Metabolic syndrome; Metformin; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Agave inulin + Metformin (Experimental): 5 g of Agave inulin powder every 12 hrs + 500 mg tablet of metformin every 24 hrs
  Interventions: Drug: Metformin; Dietary Supplement: Agave inulin
- Metformin + Placebo of agave inulin (Active Comparator): 500 mg tablet of metformin every 24 hrs + 5 g every 12 hrs of calcinated magnesia powder
  Interventions: Drug: Metformin; Other: Placebo of agave inulin
- Agave Inulin+Placebo of Metformin (Active Comparator): 5 g of agave inulin powder every 12 hrs + 500 mg tablet of calcinated magnesia as metformin placebo every 24 hrs
  Interventions: Dietary Supplement: Agave inulin; Other: Metformin placebo
- Placebo of Inulin + Placebo of Metformin (Placebo Comparator): 5 g of calcinated magnesia powder every 12 hrs + 500 mg tablet of calcinated magnesia every 24 hrs
  Interventions: Other: Placebo of agave inulin; Other: Metformin placebo

INTERVENTIONS:
Drug: Metformin — Metformin in tablet presentation of 500 mg
  Other Names: GLUCOPHAGE
  Arms: Agave inulin + Metformin; Metformin + Placebo of agave inulin
Dietary Supplement: Agave inulin — Inulin in powder obtained from agave plant, it was given to each patient a full 10 mg container.
  Arms: Agave Inulin+Placebo of Metformin; Agave inulin + Metformin
Other: Placebo of agave inulin — Calcinated magnesia powder
  Arms: Metformin + Placebo of agave inulin; Placebo of Inulin + Placebo of Metformin
Other: Metformin placebo — Calcinated magnesia tablet
  Arms: Agave Inulin+Placebo of Metformin; Placebo of Inulin + Placebo of Metformin

SUMMARY:
Presence of metabolic syndrome (MetS) and its relation with insulin resistance, obesity, dyslipidemia, systemic inflammation and cardiovascular disease is of great concern. The study of certain adipokines such as adiponectin has demonstrated an inverse association with insulin resistance, especially in Latin population lower levels of adiponectin have been observed compared to other ethnic groups. It appears to be an important molecule that is involved in limiting the pathogenesis of obesity-linked disorders and may have potential benefits as a marker to evaluate the effect of possible interventions on the MetS components and its complications.

Metformin is treatment of choice in patients with MetS, due to its low cost and pharmacological comparable effects with thiazolidinediones (pioglitazone), it decreases hyperinsulinemia, insulin resistance, free fatty acids and triglycerides, it produces as well, a moderate weight loss, improves lipid profile and delays the appearance of diabetes mellitus in subjects with an abnormal fasting glucose.

A second choice to lower the risks would be the addition of a fiber like inulin, a prebiotic, since it has demonstrated metabolic benefits on lipid and carbohydrates metabolism by several mechanisms proposed such as induction of lipogenic enzymes by glucose, production of short-chained fatty acids, glucose-dependent insulinotropic peptide (GIP) and glucagon-like peptide-1 (GLP-1), and growth of Bifidobacterium. A good natural source of inulin is the agave.

It is expected that the combination of metformin plus agave inulin will produce a beneficial impact through pharmacological synergism and that will produce changes in the pathophysiology of MetS.

DETAILED DESCRIPTION:
The main objective was to compare the effect of the administration of Metformin/agave inulin vs. Agave inulin on adiponectin in patients with MetS. The investigators conducted a double-blinded randomized trial, on 4 groups, each group with 10 male patients of 40-80 years of age with METS diagnosed by International Diabetes Federation (IDF) criteria. Randomization determined the group assignation during the 12-week trial, each group consisted of:

Group (A) Metformin plus agave inulin: 10 individuals received metformin in a dosis of 500 mg per day (1 tablet of 500 mg) plus inulin in a dosis of 10 mg per day (5 mg every 12 hours) during 12 weeks.

Group (B) Metformin plus Placebo of agave inulin: 10 individuals received Metformin in a dosis of 500mg per day (with the first bite of the second meal) plus homologue placebo of inulin (calcinated magnesia) in a dosis of 10 mg every 24 hrs (5 mg of calcinated magnesia powder every 12 hours) during 12 weeks.

Group (C) Agave inulin plus Placebo of Metformin: 10 individuals received inulin in a dosis of 10 mg every 24 hrs (5 mg every 12 hours) plus homologate placebo of metformin (calcinated magnesia) in a dosis of 500 mg per day (with the first bite of the second meal) during 12 weeks.

Group (D) Placebo of Agave inulin plus Placebo of Metformin: homologate placebo of Inulin (calcinated magnesia powder) in a dosis of 10 mg every 24 hrs (5 mg every 12 hours) plus homologate placebo of metformin (calcinated magnesia capsules) in a dosis of 500 mg per day (with the first bite of the second meal) during 12 weeks.

The clinical findings and laboratory test included a metabolic profile and biosafety, which was determined at baseline and at 12 weeks.

Waist, body weight, body fat, body mass index (BMI) and blood pressure were determined at baseline, follow up and final visit, likewise, a blood sample was obtained, centrifuged and stored at -80° degrees Celsius to be analyzed after within 30 days. The investigators assessed glucose, total cholesterol, c-HDL, c-LDL, triglycerides by enzymatic techniques, and adiponectin and insulin by ELISA. Insulin resistance (IR) was estimated by the homeostasis model assessment (HOMA) with the formula for the HOMA (fasting insulin mcg/L x (fasting glucose (mmol/L)/22.5) Adverse events and adherence to treatment were documented every 4 weeks.

Statistical analysis: Values were expressed as mean and standard deviation. Mann-Whitney U Test, Wilcoxon exact test and Kruskal-Wallis. A statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metabolic syndrome by IDF criteria

  * a person to be defined as having the metabolic syndrome they must have: Central obesity (defined as waist circumference* with ethnicity specific values) ≥80 cm in females and ≥90 cm in males; and plus any two of the following four factors:
  * Raised triglycerides ≥ 150 mg/dL (1.7 mmol/L) or specific treatment for this lipid abnormality Reduced HDL cholesterol
  * < 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females or specific treatment for this lipid abnormality
  * Raised blood pressure systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg or treatment of previously diagnosed hypertension
  * Raised fasting plasma glucose (FPG) ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes
* Age ranging from 40 to 80 years old
* Male patients
* Informed written consent

Exclusion Criteria:

* Kidney disease
* Hepatic disease
* Thyroid disease
* Diabetes mellitus
* Ischemic heart disease
* Drug consumption
* Alcohol consumption of more than 2 ounces daily
* Consumption of drugs that intervene with lipid or glucose metabolism 2 months before
* Blood pressure >160/100 mmHg.
* Lack of adherence to treatment (adherence <80%)

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on adiponectin levels (ng/mL) at 12 weeks | 12 weeks
  Before and after intervention determination of adiponectin using ELISA following the suppliers recommendations

SECONDARY OUTCOMES:
Change from Baseline in Fasting plasma glucose at 12 weeks | 12 weeks
  Before and after intervention by glucose oxidase
Change from Baseline in Total cholesterol at 12 weeks | 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Triglycerides at 12 weeks | 12 weeks
  Before and after intervention by spectrophotometry
Change from baseline in High-density lipoprotein cholesterol at 12 weeks | 12 weeks
  Before and after intervention by spectrophotometry
Changes of Insulin levels from baseline to 12 weeks | 12 weeks
  Before and after intervention by ELISA
Change of HOMA-IR from base line to 12 weeks | 12 weeks
  Before and after intervention by using the formula for the homeostasis model assessment index (FI x (fasting glucose (mmol/l)/22.5)
Change of waist circumference | 12 weeks
  Measured with a non elastic tape at baseline and after intervention
Change of body mass index | 12 weeks
  before and after intervention using a tetrapolar bioelectrical impedance analyzer (body composition analyzer
Change from baseline in Peripheral systolic blood pressure | 12 weeks
  Before and after intervention using a digital sphygmomanometer
Change from baseline in Peripheral diastolic blood pressure | 12 weeks
  Before and after intervention using a digital sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Grover, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Universidad de Guadalajara, Guadalajara, Jalisco, México, Mexico

IPD SHARING:
Plan to Share IPD: No